CLINICAL TRIAL: NCT01862185
Title: Pengaruh Pemeriksaan Procalcitonin Semikuantitatif Terhadap Adekuasi Terapi Antibiotik Empirik Awal Dan Mortalitas Pada Pasien Sepsis
Brief Title: The Effect of Semi-quantitative Procalcitonin Assay to The Adequacy of Empirical Antibiotics and Mortality in Septic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dana Dharaniyadewi, student, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: AB-PCTQ1
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Sepsis
Keywords: semiquantitative; procalcitonin; sepsis; antibiotics; mortality
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- semi-quantitative procalcitonin (Experimental): patients whom checked semi-quantitative procalcitonin examination
  Interventions: Other: semi-quantitative procalcitonin
- control (No Intervention): patients whom do not checked semi-quantitative procalcitonin examination

INTERVENTIONS:
Other: semi-quantitative procalcitonin
  Other Names: PCT-Q
  Arms: semi-quantitative procalcitonin

SUMMARY:
Sepsis is a serious clinical condition with a considerable morbidity and mortality. Procalcitonin (PCT) is a good biomarker for early diagnosis and infection monitoring. The present study aimed to investigate the effect of semi-quantitative PCT test to the empirical antibiotic initiation time, the appropriateness of empirical antibiotics and mortality in septic patients.

The hypothesis of the study are :

* There is an effect on mortality between septic patients who do and do not do semi-quantitative PCT examination
* There is an effect on empirical antibiotic initiation time between septic patients who do and do not do semi-quantitative PCT examination
* There is an effect on appropriateness of empirical antibiotic between septic patients who do and do not do semi-quantitative PCT examination

Study design is randomized diagnostic trial which is also a pragmatic trial.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years old
* have at least two concomitant systemic inflammatory response syndrome criteria
* have focal infection
* with or without sign of organ hypoperfusion or dysfunction

Exclusion Criteria:

* post operative patient
* trauma patient
* have obtained prior antibiotic
* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
mortality rate | 14 days
  mortality in 14 days since the patients were included in this study

SECONDARY OUTCOMES:
the timing of empirical antibiotic first dose | in 24 hours since the patient was diagnosis as sepsis
  when does the patient get their first dose of empirical antibiotic in 24 hours since the patient was diagnosis as sepsis?
the appropriateness of empirical antibiotic | in 24 hours since the patient was diagnosed as sepsis
  does the empirical antibiotic that given in 24 hours since the patient was diagnosis as sepsis is effective?

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dharaniyadewi, MD, Principal Investigator — Faculty of Medicine, Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia